CLINICAL TRIAL: NCT01888718
Title: Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover, Oral Bioequivalence Study of Fexofenadine Hydrochloride Orally Disintegrating Tablets 30 mg of Dr. Reddy's Laboratories Limited, India Comparing With That of Allegra ® (Containing Fexofenadine Hydrochloride) Orally Disintegrating Tablets 30 mg of Sanofi - Aventis U.S. LLC, Bridgewater, NJ 08807 in Healthy, Adult, Human Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Fexofenadine Hydrochloride Orally Disintegrated Tablets 30 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 671/10
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
MeSH Terms: interventions — fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fexofenadine Hydrochloride Orally Disintegrating (Experimental): Fexofenadine Hydrochloride Orally Disintegrating Tablets 30 mg of Dr.Reddy's Laboratories Ltd
  Interventions: Drug: Fexofenadine Hydrochloride
- ALLEGRA (Active Comparator): ALLEGRA orally disintegrating tablets 30 mg of Sanofi Aventis
  Interventions: Drug: Fexofenadine Hydrochloride

INTERVENTIONS:
Drug: Fexofenadine Hydrochloride — Fexofenadine Hydrochloride Orally Disintegrating Tablets 30 mg
  Other Names: ALLEGRA

SUMMARY:
To assess the bioequivalence of Fexofenadine Hydrochloride Orally Disintegrating Tablets 30 mg of Dr. Reddy's Laboratories Limited, India comparing with that of Allegra® (containing fexofenadine hydrochloride) Orally Disintegrating Tablets 30 mg of Sanofi - aventis U.S. LLC, Bridgewater, NJ 08807 in healthy, adult, human subjects under fasting conditions. To monitor adverse events and ensure the safety of subjects.

DETAILED DESCRIPTION:
An open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover, Oral Bioequivalence Study of Fexofenadine Hydrochloride Orally Disintegrating Tablets 30 mg of Dr. Reddy's Laboratories Limited, India Comparing With That of Allegra ® (Containing Fexofenadine Hydrochloride) Orally Disintegrating Tablets 30 mg of Sanofi - Aventis U.S. LLC, Bridgewater, NJ 08807 in Healthy, Adult, Human Subjects Under Fasting Conditions.

ELIGIBILITY:
Inclusion Criteria:

i. Provide written informed consent.

ii. Must be healthy, adult, human beings within 18 and 45 years of age (both inclusive) weighing at least 50 kg.

iii. Having a body mass index between 18.5 and 24.9 (both inclusive), calculated as weight in Kg/height in m2.

iv. Must be of normal health as determined by medical history, physical examination and laboratory investigation performed within 28 days prior to the commencement of the study. (Laboratory values must be within normal limits or considered by the physician / investigator to be of no clinical significance).

v. Female Subjects

* of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
* surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)

Exclusion Criteria

i.Incapable of understanding the informed consent.

ii. Systolic blood pressure less than 90 mm of Hg or more than 140 mm of Hg.

iii. Diastolic blood pressure less than 60 mm of Hg or more than 90 mm of Hg.

iv. Oral temperature is below 95.0°F or above 98.6°F.

v. Pulse rate below 50/min or above 100/min.

vi. History of hypersensitivity or idiosyncratic reaction to investigational drug product or any other related drugs.

vii. Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function.

viii. Consumption of grapefruit for the past ten days prior to the check-in, in each period.

ix. Regular smoker who has a habit of smoking more than nine cigarettes per day and has difficulty in abstaining from smoking during sample collection period.

x. Habit of tobacco chewing.

xi. Habit of alcoholism and difficulty in abstaining from alcohol during the sample collection period.

xii. Difficulty in abstaining from xanthine containing food or beverages (like tea, coffee, chocolates and cola drinks) during the sample collection period.

xiii. Intake of over the counter (OTC) or prescribed medications and enzyme modifying medication or systemic medication for the last 30 days before dosing.

xiv. Clinically significant abnormalities and / or with significant diseases. xv. Confirmed positive in alcohol screening.

xvi. Confirmed positive in selected drug of abuse.

xvii. Participated in any other clinical investigation using experimental drug/donated blood in past 90 days before the date of start of study.

xviii. Confirmed positive in urine pregnancy test.

xix. Female detected to be pregnant, breast feeding or who is likely to become pregnant during the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-02; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | Pre-dose (0.0) and 0.167, 0.33, 0.50, 0.75, 1.25, 1.5, 1.75, 2, 2.33, 2.67, 3, 3.50, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Vimal Teja, MD, Principal Investigator — Bioserve Clinical Research Private Limited
Locations (1):
- Bioserve Clinical Research Private Limited, Bālānagar, Hyderabad, Andhra Pradesh, India